CLINICAL TRIAL: NCT03671369
Title: Post-marketing Surveillance of GlaxoSmithKline (GSK) Biologicals' Human Papillomavirus (HPV)-16/18 Vaccine, Cervarix When Administered According to the Approved Prescribing Information in Korea
Brief Title: A Post-marketing Surveillance Study to Assess the Safety of Cervarix (GlaxoSmithKline [GSK] Biologicals' Human Papillomavirus [HPV] -16/18 Vaccine), When Administered According to the Approved Prescribing Information (PI) in Korea
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 208710
Record Dates: First submitted 2018-08-30; First posted 2018-09-14 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2022-05

CONDITIONS: Neoplasms, Rectal
Keywords: Human Papillomavirus Vaccine; Adverse events after vaccination; Safety; Serious adverse events after vaccination
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervarix Group: The study group comprised of 9-25 year-old male and female subjects who were administered with 3 doses of Cervarix vaccine, according to a 0, 1, and 6 months schedule, as per locally approved prescribing information (PI) in Korea. The 9-14 years old subjects were vaccinated with 2 doses, according to a 0 and 6-12 months schedule. In the 2-dose schedule, if the second dose was administered before 5 months after the first dose, the third dose vaccination was required. In the 3 doses schedule, if the vaccination schedule required flexibility, the second dose was administered between 1 and 2.5 months and the third dose was administered between 5 and 12 months after the first dose.
  Interventions: Other: Safety data collection (following routine vaccination) by a continuous surveillance method.

INTERVENTIONS:
Other: Safety data collection (following routine vaccination) by a continuous surveillance method. — This study assesses the safety of GSK Biologicals' Human papillomavirus (HPV) vaccine in terms of frequency and intensity of adverse events (AEs) and serious adverse events (SAEs) when administered routinely in male and female subjects aged between 9 and 25 years, according to the approved Prescribing Information in Korea.
  All AEs reported during the 30-day post-vaccination follow-up period (Day 1 to Day 30) and all SAEs reported through the study period from dose 1 up to 30 days after the last dose administered during the post-marketing surveillance (PMS) were collected as part of safety data in this PMS.

SUMMARY:
The purpose of this post-marketing surveillance (PMS) study is to collect safety information on the use of Cervarix upon the expanded indication to anal cancer to both women and men (at least 600 Korean women and men) within 30 days after each vaccination dose, when administered according to the approved prescribing information (PI) in Korea in a real health care setting over a period of 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject or/and subjects whose parent(s)/Legally Acceptable Representative(s) [LAR(s)], in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Korean male or female subjects aged 9-25 years who are eligible for the series of Cervarix according to the locally approved PI.
* Written informed consent obtained from the subject/from the parent(s)/LAR of the subject.

Exclusion Criteria:

* At the time of PMS entry, the contraindications and precautions of use indicated in the locally approved PI. PI should be checked and the subject must not be included in the PMS if there is any contraindication. Any changes in the locally approved PI must be implemented immediately.
* Subjects who had previous administration of a HPV vaccine other than Cervarix will not be enrolled into the study.
* Subjects who are not eligible for vaccination with Cervarix according to the medical judgement of physician.
* Child in care.

Ages: 9 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Korean male and female subjects aged 9-25 years, who are eligible for the series of Cervarix vaccination, according to the locally approved PI.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- South Korea (14):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Chungcheongnam-do
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gongju-si, Chungcheongnam-do
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Gyeongsangbuk-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeollabuk-do
  - GSK Investigational Site, Jeonju-si, Jeollabuk-do
  - GSK Investigational Site, Jeonju-si,Jeollabuk-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
  - GSK Investigational Site, Yangju-si, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eun BW, Bahar E, Xavier S, Kim H, Borys D. Post-marketing surveillance study of the safety of the HPV-16/18 vaccine in Korea (2017-2021). Hum Vaccin Immunother. 2023 Dec 31;19(1):2184756. doi: 10.1080/21645515.2023.2184756. Epub 2023 Mar 10. PMID 36896702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 29 centers in Republic of Korea.
Pre-assignment Details: Out of 670 subjects enrolled in the study, 1 subject did not receive any vaccine and therefore was not included in any analysis.
Period: Overall Study
Arm/Group | Cervarix Group
Started | 669
Completed | 378
Not Completed | 291
Not completed — Other | 1
Not completed — Withdrawal by Subject | 289
Not completed — Not willing to be vaccinated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cervarix Group
Number analyzed (Participants) | 669
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.92 (2.75)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23
  Female | 646
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 664
  Non-Korean | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Subjects With Adverse Events (AEs) Post Dose 1
Description: An adverse event (AE) is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. The percentage of subjects with AEs was calculated by dividing the number of subjects with adverse events by the number of subjects in each total number of Cervarix doses vaccinated in Total Safety Cohort, and multiplied by 100.
Time Frame: From Day 1 up to 30 days (post dose 1 vaccination)
Population: The analysis was performed on Total Safety cohort, which included all subjects with data available at the specified time point who received at least one dose of vaccine as per the protocol and who reported adverse events even though they have not completed 30-days follow-up period after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 457
Percentage of subjects | 17.72 [14.33 to 21.54]

2. Primary Outcome: Percentage (%) of Subjects With Adverse Events (AEs) Post Dose 2
Description: as for outcome 1
Time Frame: From Day 1 up to 30 days (post dose 2 vaccination)
Population: The analysis was performed on Total Safety cohort, which included all subjects with data available at the specified time point who received two doses of vaccine as per the protocol and who reported adverse events even though they have not completed 30-days follow-up period after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 389
Percentage of subjects | 18.77 [15.01 to 23.01]

3. Primary Outcome: Percentage (%) of Subjects With Adverse Events (AEs) Post Dose 3
Description: as for outcome 1
Time Frame: From Day 1 up to 30 days (post dose 3 vaccination)
Population: The analysis was performed on Total Safety cohort, which included all subjects with data available at the specified time point who received three doses of vaccine as per the protocol and who reported adverse events even though they have not completed 30-days follow-up period after vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Cervarix Group
Number analyzed (Participants) | 35
Percentage of subjects | 2.86 [0.07 to 14.92]

4. Primary Outcome: Number of Participants With AEs by Maximum Intensity Post Dose 1
Description: An AE with maximum intensity are equivalent to severe AEs category (AEs which prevented normal everyday activities in a young child. Such an AE would, for example, prevent attendance at school/kindergarten/a day-care centre and can cause the parent(s)/Legally Acceptable Representative(s) to seek medical advice). The physician assessed the maximum intensity that occurred over the duration of the event for all AEs recorded during the PMS. The assessment was based on the physician's clinical judgement.
Time Frame: From Day 1 up to 30 days (post dose 1 vaccination)
Population: The analysis was performed on Total Safety cohort, which included all participants with data available at the specified time point who received at least one dose of vaccine as per the protocol and who reported adverse events even though they have not completed 30-days follow-up period after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 457
Participants | 0

5. Primary Outcome: Number of Participants With AEs by Maximum Intensity Post Dose 2
Description: as for outcome 4
Time Frame: From Day 1 up to 30 days (post dose 2 vaccination)
Population: The analysis was performed on Total Safety cohort, which included all participants with data available at the specified time point who received two doses of vaccine as per the protocol and who reported adverse events even though they have not completed 30-days follow-up period after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 389
Participants | 0

6. Primary Outcome: Number of Participants With AEs by Maximum Intensity Post Dose 3
Description: as for outcome 4
Time Frame: From Day 1 up to 30 days (post dose 3 vaccination)
Population: The analysis was performed on Total Safety cohort, which included all participants with data available at the specified time point who received three doses of vaccine as per the protocol and who reported adverse events even though they have not completed 30-days follow-up period after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 35
Participants | 0

7. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Fatal SAEs
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity, or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 to 30 days after the last vaccine dose administered (at Month 0 or Month 2 or Month 6)
Population: The analysis was performed on the Total Safety cohort, which included all participants who received at least one dose of vaccine as per the protocol and who reported adverse events even though they have not completed 30 days follow up period after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group
Number analyzed (Participants) | 662
Participants
  Serious Adverse Events | 0
  Fatal Serious Adverse Events | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events: From Day 1 up to 30 days (post dose 1, dose 2 and dose 3 vaccination). SAEs: From Day 1 to 30 days after the last vaccine dose administered (at Month 0 or Month 2 or Month 6).
Description: Data was collected based on the Total Vaccinated Cohort.
Arm/Group | Cervarix Group
All-Cause Mortality (participants affected / at risk) | 0/669
Serious Adverse Events (participants affected / at risk) | 0/669
Other Adverse Events (participants affected / at risk) | 144/669
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=669)
Injection site pain (General disorders) | 60 (68)
Injection site erythema (General disorders) | 31 (34)
Injection site swelling (General disorders) | 13 (13)
Pyrexia (General disorders) | 12 (12)
Injection site pruritus (General disorders) | 4 (4)
Injection site bruising (General disorders) | 2 (2)
Injection site paraesthesia (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Injection site oedema (General disorders) | 1 (1)
Injection site rash (General disorders) | 1 (1)
Injection site warmth (General disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 7 (7)
Nasopharyngitis (Infections and infestations) | 5 (5)
Pharyngitis (Infections and infestations) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Chronic sinusitis (Infections and infestations) | 2 (2)
Paronychia (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 4 (4)
Syncope (Nervous system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chalazion (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Lip swelling (Immune system disorders) | 1 (1)
Swelling of eyelid (Immune system disorders) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
Statistical significance of AEs incidence proportion by baseline background factor wasn't planned in statistical analysis plan. As per Ministry of Food and Drug Safety regulation, additional analysis was done to determine what factors may affect AEs incidence in Korea routine clinical practice. Study design didn't include stratification or adjustment to account for baseline factors in analysis. Study findings are to be interpreted with caution considering clinical plausibility and significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT03671369/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03671369/SAP_001.pdf